CLINICAL TRIAL: NCT05836714
Title: Validation of a Viable Delirium Detection Test Performed by Nurses and Physicians During Routine Patient Care
Brief Title: Delirium Detection During Routine Patient Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0094-18-BNZ
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Delirium
Keywords: DELIRIUM; DIAGNOSIS; 4AT
MeSH Terms: conditions — Delirium; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the presence of validated tests, there are still drawbacks to implementing delirium diagnosis tests in hospital wards. We developed a new, simple, easy to implement user friendly delirium diagnostic test that is likely to facilitate implementation in many departments. The present study will compare the new test to a well validated older test - 4AT.

DETAILED DESCRIPTION:
Delirium is characterized by an acute onset altered mental status and/or a confusional state. Although delirium has been known since ancient times, the condition is often not diagnosed, documented, evaluated, and managed. Early detection of delirium in hospitalized patients may be critical, particularly on internal medicine wards, as mental deterioration in the elderly can be the first sign of preventable diseases and disorders that precipitate delirium. Nevertheless only 15%-35% of cases of delirium in hospitalized patients are identified by the treating staff and documented in the medical records. The main reasons for this shortcoming are insufficient awareness to emerging delirium, and excessive work load.

We have recently developed and implemented in our Department of Internal Medicine a new diagnostic tool for delirium. This test, designated R&M, is based on a combination of RADAR (Recognizing Acute Delirium As part of your Routine), performed by the nurses during medication dispensing, and MOYB (Months Of the Year Backwards), performed by residents during the routine rounds in patients with positive RADAR. Both tests are online and saved in the patients' electronic records.

The purpose of this study is to demonstrate non-inferiority of R&M compared to 4AT (Attention, Abbreviated mental test, Alertness, Acute onset Test), an old and well validated delirium recognition test. The sample size required for a sensitivity of 95% and a 95% confidence interval was calculated to be n=365, assuming delirium prevalence of >20% in elderly patients hospitalized in internal medicine wards.

ELIGIBILITY:
Inclusion Criteria:

- patients >70 yrs old, hospitalized in the department of internal medicine

Exclusion Criteria:

* severe dementia

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients >70 yrs old, hospitalized in the department of internal medicine
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Validation of a viable delirium detection test care. | ONE YEAR
  non-inferiority of a new delirium detection test (R&M) compared to 4AT.

CONTACTS AND LOCATIONS:
Overall Officials: RON OLIVEN, MD, Principal Investigator — BNAI-ZION MC HAIFA ISRAEL
Locations (1):
- Bnai-Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided